CLINICAL TRIAL: NCT01725074
Title: Koronare Herzkrankheit Projekt Mannheim
Brief Title: Randomized Control Trial to Evaluate Effectiveness of a Case Managment Program Regarding Psychosocial Well-being and Disease Symptoms Health for Patients With Multimorbid Coronary Heart Disease (CHD) Patients (KHK ProMA)
Acronym: KHK ProMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genossenschaft Gesundheitsprojekt Mannheim e.G (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); pfm medical Institute gGmbH, Germany (Unknown); Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHK ProMA
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Coronary Heart Disease; Multimorbidity
Keywords: Coronary Heart Disease, multimorbidity, primary care, case management, loneliness, depression, social support
MeSH Terms: conditions — Coronary Disease; Depression | interventions — Drug Interactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Case Management "CM CHD" (Experimental): The intervention consists of a biweekly telephone or personal contact by trained case managers over the first 6-months and monthly contact over the second 6-months to assess well-being, everyday life (positive, neutral and negative daily events), and to inquire after health and personal problems on which basis the case manager offers practical or emotional support or a referral to the general practitioner if deemed necessary. During the contacts also medical control measures like blood pressure or weight are taken, and other study outcome measures like need for medical treatment.
  Interventions: Behavioral: Case Management "CM CHD"
- Social Interaction (Experimental): Identical as the CM CHD group, but with exclusion of medical control measures.
  Interventions: Behavioral: Social Interaction
- Control Group (No Intervention): Patients assigned to the control group received usual care (no additional contact/support) and therefore stays under the standard supervision of the general practitioner i.e. as participant in the normal disease management program for CHD (quarterly check-ups).

INTERVENTIONS:
Behavioral: Case Management "CM CHD" — Patients, who are randomized to the intervention group, will receive case management from a trained and experienced physician assistant. The case manager will carry out following tasks:
  * Biweekly/monthly telephone consultations or home visits
  * Identification of health or personal problems of the patient
  * Monitoring of medical parameters
  * Coordination of contact with health care providers if necessary
  * Support to the patient related to health status and environmental changes
  * Promote disease-self management through coaching
  * Counseling, that is focused on emotional support and active listening
  Arms: Case Management "CM CHD"
Behavioral: Social Interaction — Identical as the CM CHD group, but with exclusion of medical control measures and the medical aspects.
  Arms: Social Interaction

SUMMARY:
This randomized controlled trial (RCT) will examine a case management program for patients suffering from coronary heart disease with multimorbidity in Mannheim, Germany. The trail consists of 3 treatment arms: 1) intensified case management; 2) social interaction alone 3) standard care. The main objectives are to evaluate how case management and social interaction alone compared to standard medical care affect the primary and secondary outcomes: physical health, quality of life, loneliness, depression, self-efficacy, outcome expectancies, social support, health locus of control, lifestyle behavior, social network, vulnerability, intention, severity, health worries and cognitive functions.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) will examine a case management program for 320 male and female patients suffering from coronary heart disease with multimorbidity in Mannheim, Germany. The main objectives are to evaluate how case management and social interaction alone compared to standard medical care affect the primary and secondary outcomes: physical health, quality of life, loneliness, depression, self-efficacy, outcome expectancies, social support, health locus of control, lifestyle behavior, social network, vulnerability, intention, severity, health worries and cognitive functions.

Additionally, the secondary outcomes are studied as factors that mediate the effects of case management and social interaction alone compared to standard medical care on the primary outcomes.

The trail consists of 3 treatment arms: 1) intensified case management; 2) social interaction alone 3) usual care. The intervention consists of a biweekly contact by trained case managers over the first 6-months and a monthly contact over the subsequent 6-months. Each contact involves an assessment of well-being, daily life, problems and offering emotional support and solutions or refer to the general practitioner if necessary (both intervention groups).

For patients assigned to the "CM CHD" the contacts include medical control (like blood pressure or weight) and well-being as well as an additional core set of relevant outcome measures (e.g. need for treatment of fatigue).

Patients assigned to the control group received usual care (no CM or contact). An additional fourth group is monitored. This group is consisting of patients who refused to take part in the study but gave consent to collect their practice data (not randomized).

Each patient will be followed for 12 months. Extensive assessments and self-administered questionnaires take place at baseline, 6-month and 12-month for all patients in the three randomized groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed CHD

  * participation in the Disease Management Program (DMP) of CHD or
  * a risk score (Framingham or Procam) higher than 20%
* two additional chronic diseases (multimorbid)

Exclusion Criteria:

* Patients living in institutionalized care
* Patients having dementia
* Patients associated with a life expectancy of less than one year
* Patients who are not able to communicate in German language

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Change in health outcomes | Measured at baseline, 6 and 12 months follow-up
  This includes biomarkers (blood pressure, BMI, weight, blood lipids), physical balance performance (semi tandem stand), care utilization and medication usage, clinical assessments and need for (medical) treatment (like dyspnea, fatigue, care, vomitus, thirst, lack of appetite, nausea, disorientation).
  Within the intervention group CM CHD weight and blood pressure is self-reported by patients biweekly within the first six months and monthly within the second six months.
Change in quality of life | Measured at baseline, 6 and 12 months follow-up
  We will measure this variable using the "EQ-5D" and two additional items.

SECONDARY OUTCOMES:
Change in Loneliness | Measured at baseline, 6 and 12 months follow-up
  We will measure this variable using the "Hamburger Einsamkeits-Skala (HES)" a German version of the UCLA-Loneliness Scale.
Change in Depression | Measured at baseline, 6 and 12 months follow-up
  We will measure this variable using the "Patient Health Questionnaire - 9 item (PHQ-9) instrument".
Change in self-efficacy | Measured at baseline, 6 and 12 months follow-up
  We will measure this variable using the "SWE" questionnaire as well as items of self-efficacy regarding sports, quit smoking and healthier eating behavior.
Change in social support | Measured at baseline, 6 and 12 months follow-up
  We will measure this variable using the "Skala sozialer Unterstützung bei Krankheit (SSUK)". This instrument consists of two subscales, supportive behavior as well as stressful interactions.
Change in health locus of control | Measured at baseline, 6 and 12 months follow-up
  We will measure this variable using the "MHLC-C". This instrument consists of four subscales, internal, chance, doctors and other people.
Change in lifestyle behavior | Measured at baseline, 6 and 12 months follow-up
  This includes smoking, alcohol consumption, eating habits and physical activity.
Change in social network of family and friends | Measured at baseline, 6 and 12 months follow-up
  This includes the number of closer family members and friends and the amount of contact with them.
Change in outcome expectancies | Measured at baseline, 6 and 12 months follow-up
  This includes items regarding sports, quit smoking and healthier eating behavior.
Change in vulnerability | Measured at baseline, 6 and 12 months follow-up
  This includes the total vulnerability regarding specific diseases for one's own person as well as for a peer/other person. Thus the relative vulnerability can be determined.
Change in intention | Measured at baseline, 6 and 12 months follow-up
  This includes items of intentions for a healthier lifestyle like more physical activity, quit smoking and healthier eating behaviors.
Change in severity | Measured at baseline, 6 and 12 months follow-up
  This includes the estimated severity of different cardiovascular diseases in general as well as their severity for the own individual.
Change in health worries | Measured at baseline, 6 and 12 months follow-up
  This includes worries about the own health in general as well as regarding specific health problems like blood pressure, high cholesterol or the risk of a myocardial infarction.
Change in cognitive functions | Measured at baseline, 6 and 12 months follow-up
  This will be measured using the Mini-mental Status Exam and the Clock Drawing Test.

CONTACTS AND LOCATIONS:
Locations (1):
- Genossenschaft Gesundheitsprojekt Mannheim e.G., Mannheim, Baden-Wurttemberg, Germany